CLINICAL TRIAL: NCT05977296
Title: The Effects of Continuous Positive Airway Pressure (CPAP) on Oral Frailty and Dysphagia in Patients With Obstructive Sleep Apnea(OSA): A Prospective Cohort Study Design
Brief Title: Obstructive Sleep Apnea (OSA), Oral Frailty, Dysphagia, Continuous Positive Airway Pressure (CPAP)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Chen, Yen-Chin, Vice Head Nurse and Clinical Assistant Professor, National Cheng-Kung University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A-ER110-551
Record Dates: First submitted 2023-07-18; First posted 2023-08-04 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2024-08

CONDITIONS: Dysphagia; OSA; CPAP
Keywords: Obstructive sleep apnea; Oral frailty; Dysphagia; CPAP
MeSH Terms: conditions — Deglutition Disorders; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- OSA patients (Experimental): The experimental group in this study consisted of individuals who were assigned to the CPAP (Continuous Positive Airway Pressure) intervention. Participants in the experimental group were instructed to wear a CPAP device during their sleep.
  Interventions: Device: CPAP
- Usual group (No Intervention): In the control group, participants received standard or routine nursing care without any specific interventions(CPAP) or modifications. The standard nursing care provided to the participants followed established protocols and guidelines commonly practiced in general healthcare settings.

INTERVENTIONS:
Device: CPAP — To use CPAP
  Arms: OSA patients

SUMMARY:
The purpose of this study is to evaluate the effects of the CPAP treatment on oral frailty and dysphagia among OSA patients.

DETAILED DESCRIPTION:
The research will be divided into three stages. The first stage will investigate the incidence of OSA in patients over 50 years old using the National Health Insurance Research Database (NHIRD). The second stage will examine the relationships among OSA, oral frailty, and dysphagia through an observational case-control study with 225 OSA patients and 225 controls. The third stage will evaluate the effects of CPAP treatment on oral frailty and dysphagia among moderate-severe OSA persons through a prospective cohort study with repeat four times measurements.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 years or older.
* Medically diagnosed with obstructive sleep apnea (apnea and hypopnea index, AHI, ≥ 5 events per hour).
* Clear consciousness and able to communicate in Mandarin or Taiwanese.

Exclusion Criteria:

* Central sleep apnea patients.
* Patients with neurological or muscular disorders (such as stroke or Parkinson's disease).
* Patients diagnosed with oral cancer currently undergoing oral treatment.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2022-04-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Baseline_Poor occlusal force | Baseline
  The investigators will determine the total count of natural teeth and fixed dentures among the participants. If the combined number of natural teeth and fixed dentures is below 20, it indicates a reduced occlusal force.
Within 1-month_Poor occlusal force | 2 or 4 weeks, 3 months, 6 months
  The investigators will determine the total count of natural teeth and fixed dentures among the participants. If the combined number of natural teeth and fixed dentures is below 20, it indicates a reduced occlusal force.
3-month_Poor occlusal force | 3 months
  The investigators will determine the total count of natural teeth and fixed dentures among the participants. If the combined number of natural teeth and fixed dentures is below 20, it indicates a reduced occlusal force.
6-month_Poor occlusal force | 6 months
  The investigators will determine the total count of natural teeth and fixed dentures among the participants. If the combined number of natural teeth and fixed dentures is below 20, it indicates a reduced occlusal force.
Baseline_Poor masticatory function | Baseline
  The investigators will utilize a 14-food group questionnaire to evaluate the masticatory function of the participants. If participants select 'difficult to eat' as their response for four items, it indicates a decline in the masticatory function.
Within 1-month_Poor masticatory function | 2 or 4 weeks
  The investigators will utilize a 14-food group questionnaire to evaluate the masticatory function of the participants. If participants select 'difficult to eat' as their response for four items, it indicates a decline in the masticatory function.
3-month_Poor masticatory function | 3 months
  The investigators will utilize a 14-food group questionnaire to evaluate the masticatory function of the participants. If participants select 'difficult to eat' as their response for four items, it indicates a decline in the masticatory function.
6-month_Poor masticatory function | 6 months
  The investigators will utilize a 14-food group questionnaire to evaluate the masticatory function of the participants. If participants select 'difficult to eat' as their response for four items, it indicates a decline in the masticatory function.
Baseline_Poor tongue-lip motor function | Baseline
  The investigators will assess the oral-diadochokinesis of the participants. Each participant will be instructed to repeat the syllables /pa/, /ta/, and /ka/ for a duration of 5 seconds. If the number of /pa/ syllables produced per second is below 6, it indicates a decline in tongue-lip motor function.
Within 1-month_Poor tongue-lip motor function | 2 or 4 weeks
  The investigators will assess the oral-diadochokinesis of the participants. Each participant will be instructed to repeat the syllables /pa/, /ta/, and /ka/ for a duration of 5 seconds. If the number of /pa/ syllables produced per second is below 6, it indicates a decline in tongue-lip motor function.
3-month_Poor tongue-lip motor function | 3 months
  The investigators will assess the oral-diadochokinesis of the participants. Each participant will be instructed to repeat the syllables /pa/, /ta/, and /ka/ for a duration of 5 seconds. If the number of /pa/ syllables produced per second is below 6, it indicates a decline in tongue-lip motor function.
6-month_Poor tongue-lip motor function | 6 months
  The investigators will assess the oral-diadochokinesis of the participants. Each participant will be instructed to repeat the syllables /pa/, /ta/, and /ka/ for a duration of 5 seconds. If the number of /pa/ syllables produced per second is below 6, it indicates a decline in tongue-lip motor function.
Baseline_Low tongue pressure | Baseline, 2 or 4 weeks, 3 months, 6 months
  The investigators will employ the YBERMEDIC Tongue Depressor, a tongue pressure measuring instrument, to assess the maximum tongue pressure. Participants will be instructed to press a balloon attached to their tongue against the anterior palate for several seconds, repeating this process three times. If the maximum tongue pressure is below 30 kPa, it indicates a decline in tongue pressure.
Within 1-month_Low tongue pressure | 2 or 4 weeks
  The investigators will employ the YBERMEDIC Tongue Depressor, a tongue pressure measuring instrument, to assess the maximum tongue pressure. Participants will be instructed to press a balloon attached to their tongue against the anterior palate for several seconds, repeating this process three times. If the maximum tongue pressure is below 30 kPa, it indicates a decline in tongue pressure.
3-month_Low tongue pressure | 3 months, 6 months
  The investigators will employ the YBERMEDIC Tongue Depressor, a tongue pressure measuring instrument, to assess the maximum tongue pressure. Participants will be instructed to press a balloon attached to their tongue against the anterior palate for several seconds, repeating this process three times. If the maximum tongue pressure is below 30 kPa, it indicates a decline in tongue pressure.
6-month_Low tongue pressure | 6 months
  The investigators will employ the YBERMEDIC Tongue Depressor, a tongue pressure measuring instrument, to assess the maximum tongue pressure. Participants will be instructed to press a balloon attached to their tongue against the anterior palate for several seconds, repeating this process three times. If the maximum tongue pressure is below 30 kPa, it indicates a decline in tongue pressure.
Baseline_Low swallowing tongue pressure | Baseline
  The investigators will employ the YBERMEDIC Tongue Depressor, a tongue pressure measuring instrument, to assess the maximum swallowing tongue pressure. Participants will be instructed to swallow their saliva, repeating this process three times. If the maximum tongue pressure is below 15.46 kPa, it indicates a decline in swallowing tongue pressure.
Within 1-month_Low swallowing tongue pressure | 2 or 4 weeks
  The investigators will employ the YBERMEDIC Tongue Depressor, a tongue pressure measuring instrument, to assess the maximum swallowing tongue pressure. Participants will be instructed to swallow their saliva, repeating this process three times. If the maximum tongue pressure is below 15.46 kPa, it indicates a decline in swallowing tongue pressure.
3-month_Low swallowing tongue pressure | 3 months
  The investigators will employ the YBERMEDIC Tongue Depressor, a tongue pressure measuring instrument, to assess the maximum swallowing tongue pressure. Participants will be instructed to swallow their saliva, repeating this process three times. If the maximum tongue pressure is below 15.46 kPa, it indicates a decline in swallowing tongue pressure.
6-month_Low swallowing tongue pressure | 6 months
  The investigators will employ the YBERMEDIC Tongue Depressor, a tongue pressure measuring instrument, to assess the maximum swallowing tongue pressure. Participants will be instructed to swallow their saliva, repeating this process three times. If the maximum tongue pressure is below 15.46 kPa, it indicates a decline in swallowing tongue pressure.
Baseline_Dysphagia | Baseline
  The investigators will use the Eating Assessment Tool (EAT-10) to evaluate participants' swallowing difficulties. The EAT-10 is a straightforward assessment consisting of 10 questions, each assigned a score ranging from 0 (none) to 4 (severe). If the EAT-10 score is 3 or higher, it indicates that participants may experience challenges in swallowing efficiently and safely
Within 1-month_Dysphagia | 2 or 4 weeks
  The investigators will use the Eating Assessment Tool (EAT-10) to evaluate participants' swallowing difficulties. The EAT-10 is a straightforward assessment consisting of 10 questions, each assigned a score ranging from 0 (none) to 4 (severe). If the EAT-10 score is 3 or higher, it indicates that participants may experience challenges in swallowing efficiently and safely
3-month_Dysphagia | 3 months
  The investigators will use the Eating Assessment Tool (EAT-10) to evaluate participants' swallowing difficulties. The EAT-10 is a straightforward assessment consisting of 10 questions, each assigned a score ranging from 0 (none) to 4 (severe). If the EAT-10 score is 3 or higher, it indicates that participants may experience challenges in swallowing efficiently and safely
6-month_Dysphagia | 6 months
  The investigators will use the Eating Assessment Tool (EAT-10) to evaluate participants' swallowing difficulties. The EAT-10 is a straightforward assessment consisting of 10 questions, each assigned a score ranging from 0 (none) to 4 (severe). If the EAT-10 score is 3 or higher, it indicates that participants may experience challenges in swallowing efficiently and safely
Baseline_Oral Health status | Baseline
  The Oral Health Assessment Tool (OHAT) is a clinical assessment tool designed for frail older individuals to self-evaluate their oral health status. It encompasses eight categories of oral health, including lips, tongue, gums and oral tissue, natural teeth, dentures, oral cleanliness, saliva secretion, and dental pain. Each category is assessed on a scale of 0 (healthy), 1 (changes), or 2 (unhealthy). The overall scores range from 0 to 16, with a higher OHAT score indicating poorer oral health.
Within 1-month_Oral Health status | 2 or 4 weeks
  The Oral Health Assessment Tool (OHAT) is a clinical assessment tool designed for frail older individuals to self-evaluate their oral health status. It encompasses eight categories of oral health, including lips, tongue, gums and oral tissue, natural teeth, dentures, oral cleanliness, saliva secretion, and dental pain. Each category is assessed on a scale of 0 (healthy), 1 (changes), or 2 (unhealthy). The overall scores range from 0 to 16, with a higher OHAT score indicating poorer oral health.
3-month_Oral Health status | 3 months
  The Oral Health Assessment Tool (OHAT) is a clinical assessment tool designed for frail older individuals to self-evaluate their oral health status. It encompasses eight categories of oral health, including lips, tongue, gums and oral tissue, natural teeth, dentures, oral cleanliness, saliva secretion, and dental pain. Each category is assessed on a scale of 0 (healthy), 1 (changes), or 2 (unhealthy). The overall scores range from 0 to 16, with a higher OHAT score indicating poorer oral health.
6-month_Oral Health status | 6 months
  The Oral Health Assessment Tool (OHAT) is a clinical assessment tool designed for frail older individuals to self-evaluate their oral health status. It encompasses eight categories of oral health, including lips, tongue, gums and oral tissue, natural teeth, dentures, oral cleanliness, saliva secretion, and dental pain. Each category is assessed on a scale of 0 (healthy), 1 (changes), or 2 (unhealthy). The overall scores range from 0 to 16, with a higher OHAT score indicating poorer oral health.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University Hospital, College of Medicine, National Cheng Kung University, Tainan, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No